CLINICAL TRIAL: NCT02860806
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Absolute Bioavailability of JNJ-63623872 Administered as an Intravenous Infusion and a 600-mg Oral Dose in Healthy Adult Subjects
Brief Title: Safety, Tolerability, Pharmacokinetic and Absolute Bioavailability Study of JNJ-63623872 Administered as an Intravenous Infusion and a 600-Milligram (mg) Oral Dose in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108196; 63623872FLZ1002 (Other: Janssen-Cilag International NV); 2016-000921-37 (EudraCT Number)
Record Dates: First submitted 2016-08-05; First posted 2016-08-09 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Healthy
MeSH Terms: interventions — pimodivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (10):
- Part 1: Period 1 (JNJ-63623872 100 mg or Placebo) (Experimental): Participants will receive a single intravenous (IV) infusion of JNJ-63623872 100 milligram (mg) [3 milligram per milliliters (mg/mL) solution] (Treatment A) or matching placebo (Treatment D) over 120 minutes.
  Interventions: Drug: JNJ-63623872; Drug: Placebo
- Part 1: Period 2 (JNJ-63623872 200 mg or Placebo) (Experimental): Participants will receive a single IV infusion of JNJ-63623872 200 mg (3 mg/mL solution) (Treatment B) or matching placebo (Treatment D) over 120 minutes.
  Interventions: Drug: JNJ-63623872; Drug: Placebo
- Part 1: Period 3 (JNJ-63623872 300 mg or Placebo) (Experimental): Participants will receive a single IV infusion of JNJ-63623872 300 mg (3 mg/mL solution) (Treatment C) or matching placebo (Treatment D) over 120 minutes.
  Interventions: Drug: JNJ-63623872; Drug: Placebo
- Part 2: Group 1 (EFG) (Experimental): Participants will receive a single IV 300-mg infusion of JNJ-63623872 (3 mg/mL solution) over x minutes (Treatment E) followed by a single IV 300-mg infusion of JNJ-63623872 (3 mg/mL solution) over y minutes (Treatment F), then a single oral 600-mg dose (2* 300 mg tablets) of JNJ-63623872 under fasted conditions (Treatment G). Study drug administration in subsequent treatment periods will be separated by a washout period of at least 7 days.
  Interventions: Drug: JNJ-63623872
- Part 2: Group 2 (FGE) (Experimental): Participants will receive Treatment F, then Treatment G followed by Treatment E. Study drug administration in subsequent treatment periods will be separated by a washout period of at least 7 days.
  Interventions: Drug: JNJ-63623872
- Part 2: Group 3 (GEF) (Experimental): Participants will receive Treatment G, then Treatment E followed by Treatment F. Study drug administration in subsequent treatment periods will be separated by a washout period of at least 7 days.
  Interventions: Drug: JNJ-63623872
- Part 2: Group 4 (GFE) (Experimental): Participants will receive Treatment G, then Treatment F, followed by Treatment E. Study drug administration in subsequent treatment periods will be separated by a washout period of at least 7 days.
  Interventions: Drug: JNJ-63623872
- Part 2: Group 5 (FEG) (Experimental): Participants will receive Treatment F, then Treatment E followed by Treatment G. Study drug administration in subsequent treatment periods will be separated by a washout period of at least 7 days.
  Interventions: Drug: JNJ-63623872
- Part 2: Group 6 (EGF) (Experimental): Participants will receive Treatment E, then Treatment G followed by Treatment F. Study drug administration in subsequent treatment periods will be separated by a washout period of at least 7 days.
  Interventions: Drug: JNJ-63623872
- Part 3: JNJ-63623872 300 mg (Experimental): Participants will receive multiple IV infusions of JNJ-63623872 300 mg (3 mg/mL) solution every 12 hours on Days 1 to 10, with only a morning dose on Day 10. Duration of infusion and dose will be selected after Part 2 of this study is completed.
  Interventions: Drug: JNJ-63623872

INTERVENTIONS:
Drug: JNJ-63623872 — 3 mg/mL solution as intravenous (IV) infusion or a single oral 600 mg dose (2 tablets of 300 mg) under fasted conditions will be administered.
Drug: Placebo — Intravenous infusion of matching placebo.
  Arms: Part 1: Period 1 (JNJ-63623872 100 mg or Placebo); Part 1: Period 2 (JNJ-63623872 200 mg or Placebo); Part 1: Period 3 (JNJ-63623872 300 mg or Placebo)

SUMMARY:
The purpose of this study is to characterize the single-dose pharmacokinetic (PK) of single escalating intravenous (IV) doses of JNJ-63623872 administered as a continuous infusion; to evaluate the safety and tolerability of single escalating IV doses of JNJ-63623872 administered as a continuous infusion; to characterize the single-dose PK of JNJ-63623872 of one selected dose administered as a continuous IV infusion at various durations and to characterize the single- and repeat-dose PK of JNJ-63623872 administered as a continuous infusion.

ELIGIBILITY:
Inclusion Criteria:

* A female participant (except if postmenopausal) must have a negative serum beta- human chorionic gonadotropin (beta-hCG) pregnancy test at screening and on Day -1 of each treatment period
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 90 days after discontinuation of study drug
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study drug, in addition to the highly effective method of contraception in the female partner, a man regardless of having been vasectomized: 1) who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (example, condom with spermicidal foam/gel/film/cream/suppository), 2) must agree not to donate sperm and 3) who is sexually active with a pregnant women must use a condom
* Must have a Body Mass Index (BMI); weight kilogram [kg]/height^2 [m]^2) between 18.0 and 30.0 kilogram per meter square (kg/m^2) (extremes included) at Screening
* Must have a blood pressure (supine after at least 5 minutes rest and standing after at least 1 minute standing) between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic at Screening

Exclusion Criteria:

* Has a history of current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* With a past history of heart arrhythmias (extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome)
* Has known allergies, hypersensitivity, or intolerance to JNJ-63623872 or its excipients
* With any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* With a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy diagnosed in previous studies with experimental drugs
* Has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening
* Has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at Screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-10 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) | Up to 10 days
  The Cmax is the maximum observed analyte concentration.
Fluctuation Index (FI) | Up to 10 days
  FI is defined as the percentage fluctuation between the Ctrough, morning analyte concentration and the maximum analyte concentration.
Average Analyte Concentration (Cavg) | Up to 10 days
  The Cavg is an average analyte concentration at steady-state over the dosing interval.
Time to Reach the Maximum Observed Analyte Concentration (Tmax) | Up to 10 days
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to 12 Hour (AUC [0-12]) | Up to 10 days
  The (AUC [0-12]) is the area under the plasma concentration-time curve from time 0 to 12 hour post dose, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC [0-last]) | Up to 10 days
  The (AUC [0-last]) is the area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Up to 10 days
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time 0 to infinity, calculated as the sum of AUC(last) and C(last)/lambda(z), where Clast is the last observed measurable (non-BQL) concentration; extrapolations of more than 20.00 percent (%) of the total AUC are reported as approximations.
Elimination Rate Constant (Lambda[z]) | Up to 10 days
  Lambda(z) is apparent terminal elimination rate constant, determined by linear regression using the terminal log-linear phase of the log transformed concentration-time curve.
Apparent Terminal Elimination Half-life (t1/2term) | Up to 10 days
  Apparent terminal elimination half-life is defined as 0.693/Lambda[z].
Systemic Clearance (CL) | Up to 10 days
  CL is the total systemic clearance, following intravenous administration.
Apparent Clearance (CL/F) | Up to 10 days
  CL/F is the total apparent clearance, following extravascular administration.
Volume of Distribution (Vd) | Up to 10 days
  The Vd is defined as volume of distribution, following single dose intravenous administration.
Apparent Volume of Distribution (Vd/F) | Up to 10 days
  Vd/F is defined as apparent volume of distribution, following single dose extravascular administration.
Volume of Distribution at Steady-State (Vss) | Up to 10 days
  Vss is defined as apparent volume of distribution at steady-state following intravenous administration.
Observed Accumulation Index (RA abs) | Up to 10 days
  Observed Accumulation Index is calculated by AUC12h, steady state/(AUC12h, single dose).
Morning Trough Analyte Concentration (Ctrough, morning) | Up to 10 days
  Ctrough, morning is defined as observed analyte concentration just prior to the beginning of a dosing interval.
Evening Trough Analyte Concentration (Ctrough, evening) | Up to 10 days
  Ctrough, evening is defined as observed analyte concentration at the end of a dosing interval.
Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to End of Study (Day 14)

SECONDARY OUTCOMES:
Absolute Bioavailability (F[abs]) | Up to 10 days
  The F(abs) is calculated as AUC (0-infinity), oral/ AUC (0-infinity), intravenous (iv)*Dose, iv/Dose, oral*100 %, where AUC (0-infinity) is area under the concentration-time curve from time zero to extrapolated infinite time, and D is the dose of administered drug.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Merksem, Belgium